CLINICAL TRIAL: NCT06718101
Title: A Phase 2 Multicenter Platform Trial of Targeted Immunomodulator Therapies for Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate the Effectiveness and Safety of Treatments, Either Alone or in Combination, for the Treatment of Moderate to Severe Atopic Dermatitis
Acronym: EMBARK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M24-727
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: Lutikizumab, ABT-981
MeSH Terms: conditions — Dermatitis, Atopic | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sub-Study 1: Lutikizumab Monotherapy (Experimental): In Period 1, participants will be receive lutikizumab Dose A at Baseline randomization, followed by Dose B every other week starting at Week 2 for 16 weeks. participants will continue into Period 2 at Week 16 with Dose C every other week until Week 52.
  Interventions: Drug: Lutikizumab
- Sub-Study 1: Placebo to Lutikizumab (Experimental): In Period 1, participants will be receive a matching placebo Dose A at Baseline randomization, followed by matching placebo Dose B every other week starting at Week 2 for 16 weeks. At Week 16, participants that were assigned placebo will then enter Period 2 and receive open-label lutikizumab Dose A , followed by lutikizumab Dose B every other week starting at Week 18, and lutikizumab Dose C every other week starting at Week 32 until Week 52.
  Interventions: Drug: Lutikizumab; Drug: Placebo

INTERVENTIONS:
Drug: Lutikizumab — Subcutaneous (SC) Injection
  Other Names: ABT-981
Drug: Placebo — Subcutaneous (SC) Injection
  Arms: Sub-Study 1: Placebo to Lutikizumab

SUMMARY:
Atopic dermatitis (AD) is a skin condition that may cause a rash and itching due to inflammation of the skin. The purpose of this study is to evaluate the clinical efficacy and safety of single therapies and/or combination therapies for moderate to severe AD through multiple substudies.

This study will consist of multiple sub-studies, Sub-Study 1 will have a randomized, placebo controlled period 1 followed by a lutikizumab treatment period 2 enrolling 80 participants at a 1 to 1 ratio.

In Sub-Study 1, participants will receive subcutaneous (SC) injections of lutikizumab or matching placebo every other week for 16 weeks followed by an additional 32 weeks of subcutaneous (SC) injections of lutikizumab every other week for a total of 52 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic and may require frequent medical assessments, blood tests, and biomarker collections.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD with onset of symptoms at least 1 year prior to the Baseline Visit and participant meets Hanifin and Rajka criteria.
* Participant has applied non-medicated, additive-free bland emollient twice daily for at least 7 days before the Baseline Visit.
* History of inadequate response to topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), or topical JAK inhibitors, OR systemic treatment for AD, OR participants for whom topical treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks).

Exclusion Criteria:

* Use of the following AD treatments within the specified washout period prior to the Baseline Visit:

  -- Systemic therapy for AD, including but not limited to corticosteroids, methotrexate, cyclosporine, azathioprine, phosphodiesterase type 4 (PDE4) inhibitors, IFN-γ, and mycophenolate mofetil within 5 half-lives [if known] or within 4 weeks, whichever is longer;

  -- Any biologic treatments, (within 5 half-lives [if known]) or within 12 weeks (whichever is longer), or as specified below: < 8 weeks for dupilumab; < 12 weeks for nemolizumab; < 16 weeks for tralokinumab and lebrikizumab.
* Phototherapy treatment, laser therapy, tanning booth, or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks.
* Herbal treatments (e.g., traditional Chinese medicines) within 4 weeks.
* Topical treatments (with the exception of non-medicated, additive-free bland emollients), including but not limited to TCS, TCIs, or topical PDE-4 inhibitors within 7 days.
* Topical JAK inhibitor within 14 days.
* Systemic JAK inhibitor (including but not limited to ruxolitinib, tofacitinib, baricitinib, upadacitinib, abrocitinib [PF-04965842], and filgotinib) within 5 half-lives [if known] or within 14 days, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving at Least a 75% Reduction in Eczema Area and Severity Index Score (EASI 75) From Baseline at Week 16 | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
Percentage of Participants Who Reported Adverse Events | Up to Week 52
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.

SECONDARY OUTCOMES:
Percentage of Participants Achieving an Improvement (Reduction) of ≥ 4 Points From Baseline in Worst Pruritus Numerical Rating Scale (WP-NRS) | At Week 4
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Percentage of Participants Achieving an EASI 50 Response | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 50 response is defined as at least a 50% reduction (improvement) from Baseline in EASI score.
Percentage of Participants Achieving an EASI 90 Response | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 90 response is defined as at least a 90% reduction (improvement) from Baseline in EASI score.
Percentage of Participants Achieving an EASI 100 Response | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for redness (erythema, inflammation), thickness (induration, papulation, swelling - acute eczema), scratching (excoriation), and lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease.
  An EASI 100 response is defined as at least a 100% reduction (improvement) from Baseline in EASI score.
Percentage of Participants Achieving an Improvement (Reduction) of ≥ 4 Points From Baseline in Worst Pruritus Numerical Rating Scale (WP-NRS) | At Week 16
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Absolute Change from Baseline for EASI | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1)] moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Percent Change From Baseline in EASI Score | At Week 16
  EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1)] moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Absolute Change from Baseline in Investigator Global Assessment for Atopic Dermatitis (vIGA-AD) | At Week 16
  The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  0 - Clear: No inflammatory signs of AD;
  1. - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
  2. - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  3. - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, oozing or crusting may be present;
  4. - Severe: Marked erythema, induration/papulation and/or lichenification; Oozing or crusting may be present.
Percentage of Participants Achieving a Validated Investigator´s Global Assessment for AD (vIGA-AD) of 0 or 1 With a Reduction From Baseline of ≥ 2 Points | At Week 16
  The vIGA-AD is a validated assessment instrument to rate the severity of atopic dermatitis globally, based on the following scale:
  * 0 - Clear: No signs of AD;
  * 1 - Almost clear: Barely perceptible erythema, induration/papulation and/or lichenification;
    - 2 - Mild: Slight but definite erythema, induration/papulation and/or minimal lichenification. No oozing or crusting;
  * 3 - Moderate: Clearly perceptible erythema, induration/papulation and/or lichenification, possible oozing or crusting;
  * 4 - Severe: Marked erythema, induration/papulation and/or lichenification; possible oozing or crusting.
Percent Change From Baseline in Worst Pruritus Numerical Rating Scale (WP-NRS) | At Week 16
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Absolute Change From Baseline in Worst Pruritus Numerical Rating Scale (WP-NRS) | At Week 16
  Participants were asked to rate itch (pruritus) intensity at its worst during the past 24 hours on a daily basis using an 11-point scale from 0 (no itch) to 10 (worst imaginable itch). Pruritus NRS was analyzed based on weekly rolling averages of daily scores.
Absolute Change from Baseline in Body Surface Area (BSA) of Atopic Dermatitis (AD) Involvement | At Week 16
  Body surface area (BSA) affected by atopic dermatitis was assessed by the physician and is expressed as a percentage of the total BSA. For purposes of the estimation, the total surface of the participant's palm plus five digits was assumed to be approximately equivalent to 1% BSA.
Percent Change from Baseline in Body Surface Area (BSA) of Atopic Dermatitis (AD) Involvement | At Week 16
  Body surface area (BSA) affected by atopic dermatitis was assessed by the physician and is expressed as a percentage of the total BSA. For purposes of the estimation, the total surface of the participant's palm plus five digits was assumed to be approximately equivalent to 1% BSA.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (30):
- United States (19):
  - Peak Dermatology Aesthetics and Wellness Fountain Hills /ID# 272550, Fountain Hills, Arizona
  - Dermatology Research Associates - Los Angeles /ID# 272945, Los Angeles, California
  - Integrative Skin Science and Research /ID# 274243, Sacramento, California
  - Clinical Trials Research Institute /ID# 274234, Thousand Oaks, California
  - Western States Clinical Res /ID# 271748, Wheat Ridge, Colorado
  - Skin Care Research Boca Raton /ID# 272544, Boca Raton, Florida
  - Research Associates of South Florida /ID# 272549, Miami, Florida
  - Advanced Clinical Research Institute /ID# 272558, Tampa, Florida
  - Encore Medical Research - Weston /ID# 272539, Weston, Florida
  - Arlington Dermatology /ID# 271735, Rolling Meadows, Illinois
  - Somnos Clinical Research /ID# 272943, Lincoln, Nebraska
  - Equity Medical, LLC /ID# 272555, New York, New York
  - Oregon Dermatology & Research Center /ID# 271733, Portland, Oregon
  - Clinical Partners /ID# 271791, Johnston, Rhode Island
  - Health Concepts /ID# 271744, Rapid City, South Dakota
  - Orion Clinical Research /ID# 274236, Austin, Texas
  - Complete Dermatology - Sugar Land /ID# 274240, Sugar Land, Texas
  - Dermatology Associates of Tyler /ID# 273684, Tyler, Texas
  - Center for Clinical Studies - Clear Lake /ID# 271749, Webster, Texas
- Japan (3):
  - Medical Corporation Kojinkai Sapporo Dermatology Clinic /ID# 273619, Sapporo, Hokkaido
  - Kyoto University Hospital /ID# 275237, Kyoto, Kyoto
  - Tachikawa Dermatology Clinic /ID# 273620, Tachikawa-shi, Tokyo
- South Korea (5):
  - Korea University Ansan Hospital /ID# 271786, Ansan-si, Gyeonggido
  - Soon Chun Hyang University Hospital Bucheon /ID# 271788, Bucheon-si, Gyeonggido
  - Seoul National University Hospital /ID# 271787, Seoul, Seoul Teugbyeolsi
  - Konkuk University Medical Center /ID# 271789, Seoul, Seoul Teugbyeolsi
  - Hallym University Kangnam Sacred Heart Hospital /ID# 271785, Seoul, Seoul Teugbyeolsi
- United Kingdom (3):
  - Royal United Hospital /ID# 274328, Bath, Bath And North East Somerset
  - Chapel Allerton Hospital /ID# 274762, Leeds, West Yorkshire
  - Royal Liverpool University Hospital /ID# 272584, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-727